CLINICAL TRIAL: NCT06484634
Title: Role of Low-Molecular-Weight Heparin in Unexplained Recurrent Pregnancy Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMWHDGKHAN
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy Loss
MeSH Terms: interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMWH Group (Experimental): Women received a daily dose of 40 mg of Low Molecular Weight Heparin subcutaneously.
  Interventions: Drug: Low molecular weight heparin
- Control (No Intervention): Women received the placebo in the form of a multivitamin tablet.

INTERVENTIONS:
Drug: Low molecular weight heparin — A daily dose of 40 mg of low-molecular-weight heparin (LMWH) subcutaneously was given to the patients.
  Arms: LMWH Group

SUMMARY:
Using low-molecular-weight heparin (LMWH), outcomes such as live birth rate and the occurrence of pregnancy complications are some of the variables reported in some studies, with varying degrees of success. The present study aimed to compare the role of LMWH in unexplained recurrent pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females between 18 and 44 years of age
* Gestational age above 8 weeks
* A history of ≥3 consecutive first trimester pregnancy losses

Exclusion Criteria:

* Patients with systemic lupus erythematosus
* Positive IgG and IgM anticardiolipin antibodies
* Positive for thrombophilia screening
* Any platelet function abnormality or a previous thromboembolic event requiring anticoagulant therapy (including heparin, aspirin or warfarin)
* Sensitive to acetylsalicylic acid, heparin, or warfarin
* Patients with any genetic, anatomical, or hormonal cause of recurrent pregnancy loss

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of Low-Molecular-Weight Heparin | 32 weeks
  Efficacy was labeled as yes in terms of live births after the age of viability, i.e., 24 weeks of gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- DG Khan Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request